CLINICAL TRIAL: NCT05047575
Title: Pilot Study of a Follow-up Intervention to Improve the Quality of Care for Low-Risk Breast Cancer Survivors
Brief Title: Remote Electronic Assessment of Survivors With Feedback Communication and Directed Referrals
Acronym: REASSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW21062; Protocol Version 12/7/2021 (Other: UW Madison); A539713 (Other: UW Madison); 2021-0961 (Other: HS-IRB UW Madison)
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
Keywords: low risk breast cancer; survivor; follow up care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REASSURE Cohort 1 (Experimental): Survivors who are enrolled at time of a follow-up visit and who will be offered the REASSURE intervention at the next 6 month visit (including the opportunity to replace a visit with feedback communication).
  Interventions: Other: REASSURE
- REASSURE Cohort 2 (Experimental): Survivors who are enrolled prior to a follow-up visit and who will be offered the REASSURE PRO assessment and feedback communication (but not provided the opportunity to replace a visit with feedback communication).
  Interventions: Other: REASSURE

INTERVENTIONS:
Other: REASSURE — REASSURE utilizes remote patient-reported outcomes assessments to comprehensively assess symptoms, promotes practice change by providing feedback reports to oncologists and engaging primary care providers (PCPs) in survivorship care, and reduces the burden of follow-up by substituting an oncology visit for thriving survivors with reassurance messaging and encouragement to pursue preventive care.
  Other Names: Remote Electronic Assessment of Survivors with Feedback Communication and Directed Referrals

SUMMARY:
This study tests a novel, risk-stratified approach for low risk breast cancer survivor follow-up care that reduces burden for survivors and their oncologists while simultaneously delivering more comprehensive care. The intervention is called Remote Electronic Assessment of Survivors with Feedback Communication and Directed Referrals (REASSURE). 50 participants will be enrolled into 2 cohorts, 25 into cohort 1 who will experience the REASSURE intervention 6 months from enrollment and 25 into cohort 2 who will experience components of the REASSURE intervention at their next follow-up visit. Participants can expect to be on study for up to 9 months.

DETAILED DESCRIPTION:
Current follow-up care for 3 million+ breast cancer survivors is both burdensome and fails to comprehensively address survivors' needs. Survivors and oncologists value these visits because visits reassure survivors about recurrence, and support oncologists' views about their responsibilities for managing ongoing therapy. However, early-stage survivors derive less benefit from follow-up, while incurring substantial financial burdens. Further, follow-up visit time restraints prevent addressing all topics prioritized by survivors or recommended as comprehensive survivorship care. Because most low-risk breast cancer survivors will never experience a recurrence, there is a critical need to develop a novel, risk-stratified approach to follow-up that reduces burden for survivors and their oncologists while simultaneously delivering more comprehensive care.

To address this gap, the team engaged stakeholders to develop an intervention for low-risk breast cancer survivors, called Remote Electronic Assessment of Survivors with Feedback Communication and Directed Referrals (REASSURE). REASSURE maintains one annual in-person oncology visit, consistent with stakeholder preferences for oncology-based follow-up. REASSURE utilizes remote patient-reported outcomes assessments to comprehensively assess symptoms, promotes practice change by providing feedback reports to oncologists and engaging primary care providers (PCPs) in survivorship care, and reduces the burden of follow-up by substituting an oncology visit for thriving survivors with reassurance messaging and encouragement to pursue preventive care. The investigators have successfully pilot tested the PRO assessment and estimate that 25% of low-risk breast cancer survivors will have symptoms requiring a follow-up visit with medical oncology.

In this pilot feasibility study, the REASSURE intervention will be implemented into clinical care for the first time. Eligible survivors will be recruited and use mixed methods to accomplish four study objectives:

* Objective 1. Assess the feasibility of implementing REASSURE into clinical practice.
* Objective 2. Determine the number of survivorship symptoms/concerns that were addressed during the follow-up visit following clinician review of the REASSURE PRO assessment.
* Objective 3. Characterize the impact of REASSURE on healthcare utilization.
* Objective 4. Assess concordance between the referral recommendation generated from the PRO assessment and medical oncologist opinion.

ELIGIBILITY:
Inclusion Criteria:

* history of stage I, ER and/or PR positive, her2neu negative breast cancer
* 12-36 months from diagnosis at the time of the survey assessment (for both REASSURE cohorts 1 and 2). For REASSURE cohort 1, this will translate into being 6-18 months from diagnosis at the time they are approached for the study.
* receiving follow-up for their breast cancer with a University of Wisconsin (UW) Breast Center medical oncologist participating in the REASSURE pilot study
* ability to complete the PRO assessment online
* English speaker

Exclusion Criteria:

* receipt of chemotherapy
* non-English speakers
* pregnancy
* cancer recurrence (local, regional or distant) since the initial diagnosis

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Feasibility: Number of Eligible Participants Enrolled | up to 6 months
  The investigator's goal is a 50% recruitment rate of eligible patients
Number of survivorship symptoms/concerns that were addressed during the follow-up visit following clinician review of the REASSURE PRO assessment | up to 9 months
  The investigator's will summarize the number of domains where survivors reported symptoms/concerns and compare that to the number of domains that were addressed, either by the PRO generated recommendation or during the follow-up visit.
Number of Participants who Replace or are Eligible to Replace a Medical Oncology Follow-Up visit with Feedback Communication | up to 1 year
  The investigator's goal is to have 33% of REASSURE cohort 1 replace a follow-up visit with medical oncology with feedback communication and REASSURE cohort 2 to be eligible to replace a follow-up visit (if the full intervention had been implemented).
Number of PRO-generated Referral Recommendations that are Concordant with Medical Oncology Opinion | up to 6 months
  The investigator's goal is to have 75% of referral recommendations be concordant with medical oncology opinion.

SECONDARY OUTCOMES:
Percent of Survivors Who Would Recommend this Approach to other survivors | up to 9 months
  Participants will be asked to answer yes or no to the following question: "Would you recommend this approach to follow-up to other survivors?"
Number of Participants Whose Concerns Were Addressed During the Preceding Visit | up to 6 months
Satisfaction with survivorship information measured with the Satisfaction with Information and Care Scale | up to 6 months
  Scored on a 5 point likert scale where 1 = very dissatisfied; 2 = dissatisfied; 3 = neutral; 4 = satisfied; 5 = very satisfied. Higher scores indicated increased satisfaction, mean score between 1-5 will be reported.
Knowledge about survivorship issues measured with the Preparing for Life as a (New) Survivor (PLANS) Scale | up to 6 months
  This is an 11 item scale, measured on a 4-point Likert scale from 0 to 3 where lower scores indicate more knowledge. Mean score between 0-3 will be reported.
Preparedness for survivorship issues measured with the Preparing for Life as a (New) Survivor (PLANS) Scale | up to 6 months
  This is a 5 item scale, measured on a 10-point Likert scale where higher scores indicate increased preparedness. Mean score between 1-10 will be reported.

OTHER OUTCOMES:
The Human Connection (THC) Scale Score | up to 9 months
  The Relationship between the survivor and oncologist (Therapeutic Alliance) will be measured using The Human Connection Scale, a 16-item questionnaire measured on a 4 point likert scale for a total possible range of scores from 16 - 64, where higher scores indicate increased therapeutic alliance.
Impact of Event Scale Score | up to 9 months
  The fear of cancer recurrence will be measured using the Impact of Event Scale, a 22-item self-report measure scored on a 5 point likert scale from 0 "not at all" to 4 "extremely", for a total possible range of scores from 0-88 where higher scores indicate increased fear of cancer recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Neuman, MD, MS, FACS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No